CLINICAL TRIAL: NCT01654419
Title: Comparison of the Quantity of Distal Movement of the Upper Canine and Molar Using Class II Elastics With and Without Sliding Jig in a Period of 3 Months
Brief Title: Comparison of the Quantity of Distal Movement of the Upper Canine and Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, LUIS ALEJANDRO SANCHEZ URIBE, PARTIAL TIME PROFESSOR IN ORTHODONTICS, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006-2010
Record Dates: First submitted 2012-07-12; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Malocclusion
Keywords: sliding jig; Class II malocclusion; Distalization mechanics; Intermaxillary elastics
MeSH Terms: conditions — Malocclusion; Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Class II elastics alone (Active Comparator): Use of class II elastics alone to correct class II dental malocclusions
  Interventions: Device: Class II elastic alone
- Class II elastics with Sliding Jig (Experimental): Class II elastics with Sliding Jig for correction of dental class II malocclusion
  Interventions: Device: Class II elastics and Sliding Jig

INTERVENTIONS:
Device: Class II elastics and Sliding Jig — Class II elastics, 3/16 6 oz, used daily for 3 months 24 hours per day and sliding jig orthodontic device
  Other Names: Archwire SS 16X22; Sliding Jig made in SS 17X25; Elastics 3/16 Heavy (6oz) Impala (Ormco)
  Arms: Class II elastics with Sliding Jig
Device: Class II elastic alone — Elastics Class II alone, used 24 hours per day for 3 months from the hook of the upper canine to the first lower molar hook
  Other Names: Elastics 3/16 heavy, 6oz. Impala (Ormco)
  Arms: Class II elastics alone

SUMMARY:
THE PURPOSE OF THE STUDY IS COMPARE THE QUANTITY OF DISTAL MOVEMENT OF THE UPPER CANINE AND MOLAR USING CLASS II ELASTICS WITH AND WITHOUT SLIDING JIG IN A PERIOD OF 3 MONTHS

DETAILED DESCRIPTION:
To achieve a Class I canine relationship at the end of the alignment and leveling phase, different intraoral devices have been used. These include intermaxillary class II elastics, which retract the upper and protract the lower arch, generating extrusive forces at the anchorage sites. Its upper distalizing action is exerted to the canine bracket and transmitted through the posterior teeth where the upper molar does not receive a direct force. The sliding jig is an auxiliary addition that exerts force to the molar by an elastic hanged in a jig between the lateral and the canine in class II; such mechanism decreases the vertical adverse effects of the elastics wearing while directing the distalizing force to the molar.

A randomized, unblinded, clinical trial comparing 30 units of analysis (hemi arches) in which were placed sliding jig or stand alone elastics were perform.

ELIGIBILITY:
Inclusion Criteria:

* Class II dental malocclusion with alignment and leveling phase ended.
* Root completed not trauma
* Second molar erupted
* Third molar absent
* Dental and periodontal health

Exclusion Criteria:

* Root uncompleted
* Dental Trauma
* Dental Pathology

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
CT analysis for comparison of distal movement of upper canine and molar using class II elastics | 3 months
  CT were taken to compare the quantity of distal movement of the upper canine and molar using class II elastics alone.

SECONDARY OUTCOMES:
CT analysis for comparison of distal movement of upper canine and molar using class II with Sliding Jig | 3 months
  CT were taken to compare the quantity of distal movement of the upper canine and molar using class II elastics with sliding jig

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Sanchez, Professor, Principal Investigator — Universidad de Antioquia
Locations (1):
- Faculty of Dentistry, Medellín, Antioquia, Colombia